CLINICAL TRIAL: NCT07163286
Title: Evaluation and Comparison of Malnutrition and Sarcopenia Risk Using PG-SGA, MUST, Nutriscore, and GLIM Criteria in Cancer Patients Undergoing Chemotherapy
Brief Title: Malnutrition and Sarcopenia Screening in Chemotherapy Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Şeyma Eroğlu, Oncology Fellowship Dr., Çanakkale Onsekiz Mart University
Other Study IDs: COMU-FNO-3
Record Dates: First submitted 2025-07-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-05

CONDITIONS: Nutrition Aspect of Cancer; Sarcopenia; Chemotherapeutic Agent Toxicity
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: The study will include approximately 150 adult outpatients diagnosed with solid tumors who are currently receiving chemotherapy. Both early and advanced stage patients of any sex aged 18 and older will be included, provided they are clinically stable and able to participate in the assessments.

SUMMARY:
The study will include approximately 150 adult outpatients diagnosed with solid tumors who are currently receiving chemotherapy. Both early and advanced stage patients of any sex aged 18 and older will be included, provided they are clinically stable and able to participate in the assessments.

DETAILED DESCRIPTION:
Background: Malnutrition and sarcopenia are prevalent and clinically significant conditions in cancer patients receiving chemotherapy. Accurate nutritional screening and early diagnosis of sarcopenia are critical for improving treatment outcomes and quality of life. Several screening tools are used for nutritional risk assessment in oncology, including PG-SGA, MUST, Nutriscore, and the recently proposed GLIM criteria.

Objective: This cross-sectional study aims to evaluate the risk of malnutrition and sarcopenia in solid tumor outpatients receiving chemotherapy. It compares the effectiveness and correlation of PG-SGA, MUST, Nutriscore, and GLIM criteria, and investigates their association with sarcopenia, measured via handgrip strength and CT-based skeletal muscle index at the L3 level.

Methods: Approximately 150 adult cancer patients receiving active outpatient chemotherapy will be assessed. Nutritional status will be evaluated using PG-SGA, MUST, Nutriscore, and GLIM. Sarcopenia will be determined via handgrip strength testing and analysis of CT images. Charlson Comorbidity Index will be used to assess comorbidity burden.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with a solid tumor (e.g., breast, lung, GI, gynecologic cancers)
* Receiving active outpatient chemotherapy
* Recent abdominal CT scan within the last 3 months or planned
* Provided written informed consent
* Physically and mentally able to complete study procedures

Exclusion Criteria:

* Declined or unable to give informed consent
* Cognitive impairment or mental status preventing participation
* Neuromuscular diseases affecting muscle mass (e.g., myopathy, MND, severe neuropathy)
* Inadequate CT image quality for L3 analysis
* Acute infection or illness within the past month
* Upper limb deformity or severe pain preventing handgrip testing
* Incomplete assessments or withdrawal of consent during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include approximately 150 adult outpatients (≥18 years) diagnosed with solid tumors (e.g., breast, lung, gastrointestinal, gynecologic cancers) who are currently receiving chemotherapy. Participants must have undergone or be scheduled for an abdominal CT scan within the last 3 months and must be physically and mentally capable of completing the assessments. Hospitalized patients and those with hematologic malignancies will be excluded.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
PG-SGA short form values | From enrollment to 6 month
Nutriscore | From enrollment to 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart University, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martin L, Birdsell L, Macdonald N, Reiman T, Clandinin MT, McCargar LJ, Murphy R, Ghosh S, Sawyer MB, Baracos VE. Cancer cachexia in the age of obesity: skeletal muscle depletion is a powerful prognostic factor, independent of body mass index. J Clin Oncol. 2013 Apr 20;31(12):1539-47. doi: 10.1200/JCO.2012.45.2722. Epub 2013 Mar 25. PMID 23530101
- [Background] Bellanti F, Lo Buglio A, Quiete S, Pellegrino G, Dobrakowski M, Kasperczyk A, Kasperczyk S, Vendemiale G. Comparison of Three Nutritional Screening Tools with the New Glim Criteria for Malnutrition and Association with Sarcopenia in Hospitalized Older Patients. J Clin Med. 2020 Jun 17;9(6):1898. doi: 10.3390/jcm9061898. PMID 32560480
- [Background] Trujillo EB, Kadakia KC, Thomson C, Zhang FF, Livinski A, Pollard K, Mattox T, Tucker A, Williams V, Walsh D, Clinton S, Grossberg A, Jensen G, Levin R, Mills J, Singh A, Smith M, Stubbins R, Wiley K, Sullivan K, Platek M, Spees CK. Malnutrition risk screening in adult oncology outpatients: An ASPEN systematic review and clinical recommendations. JPEN J Parenter Enteral Nutr. 2024 Nov;48(8):874-894. doi: 10.1002/jpen.2688. Epub 2024 Oct 16. PMID 39412097
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats A, Crivelli A, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee; GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. Clin Nutr. 2019 Feb;38(1):1-9. doi: 10.1016/j.clnu.2018.08.002. Epub 2018 Sep 3. PMID 30181091
- [Background] Arribas L, Hurtos L, Sendros MJ, Peiro I, Salleras N, Fort E, Sanchez-Migallon JM. NUTRISCORE: A new nutritional screening tool for oncological outpatients. Nutrition. 2017 Jan;33:297-303. doi: 10.1016/j.nut.2016.07.015. Epub 2016 Aug 13. PMID 27751743
- [Background] Cho JW, Youn J, Kim EM, Choi MG, Lee JE. Associations of patient-generated subjective global assessment (PG-SGA) and NUTRISCORE with survival in gastric cancer patients: timing matters, a retrospective cohort study. BMC Gastroenterol. 2022 Nov 17;22(1):468. doi: 10.1186/s12876-022-02515-3. PMID 36396994
- [Background] Baracos VE, Martin L, Korc M, Guttridge DC, Fearon KCH. Cancer-associated cachexia. Nat Rev Dis Primers. 2018 Jan 18;4:17105. doi: 10.1038/nrdp.2017.105. PMID 29345251
- [Background] Lee JS, Kim YS, Kim EY, Jin W. Prognostic significance of CT-determined sarcopenia in patients with advanced gastric cancer. PLoS One. 2018 Aug 20;13(8):e0202700. doi: 10.1371/journal.pone.0202700. eCollection 2018. PMID 30125312
- [Background] Hebuterne X, Lemarie E, Michallet M, de Montreuil CB, Schneider SM, Goldwasser F. Prevalence of malnutrition and current use of nutrition support in patients with cancer. JPEN J Parenter Enteral Nutr. 2014 Feb;38(2):196-204. doi: 10.1177/0148607113502674. PMID 24748626
- [Background] Pressoir M, Desne S, Berchery D, Rossignol G, Poiree B, Meslier M, Traversier S, Vittot M, Simon M, Gekiere JP, Meuric J, Serot F, Falewee MN, Rodrigues I, Senesse P, Vasson MP, Chelle F, Maget B, Antoun S, Bachmann P. Prevalence, risk factors and clinical implications of malnutrition in French Comprehensive Cancer Centres. Br J Cancer. 2010 Mar 16;102(6):966-71. doi: 10.1038/sj.bjc.6605578. Epub 2010 Feb 16. PMID 20160725
- [Background] Bullock AF, Patterson MJ, Paton LW, Currow DC, Johnson MJ. Malnutrition, sarcopenia and cachexia: exploring prevalence, overlap, and perceptions in older adults with cancer. Eur J Clin Nutr. 2024 Jun;78(6):486-493. doi: 10.1038/s41430-024-01433-9. Epub 2024 Apr 5. PMID 38580728